CLINICAL TRIAL: NCT02643446
Title: Serological Survey on Monitoring the Population Immunity and Positive Rate After Vaccination of Inactivated Poliovirus Vaccine
Brief Title: Serological Survey on Monitoring the Positive Rate After Vaccination of Inactivated Polio Vaccine
Acronym: IPV
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: World Health Organization (Other); Tianjin Center for Disease Control and Prevention (Unknown); Jilin Center for Disease Control and Prevention (Unknown); Hubei Provincial Center for Disease Control and Prevention (Other); Guangdong Center for Disease Prevention and Control (Other Government); Ningxia Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Huaqing Wang, Deputy Director, National Immunization Program, China CDC, Centers for Disease Control and Prevention, China
Other Study IDs: 201526
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Poliomyelitis
Keywords: Poliovirus Vaccine, Inactivated; Poliovirus Vaccine, Oral; Immunity; Seroconversion
MeSH Terms: conditions — Poliomyelitis; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (12):
- G1: IPV+OPV, 1 m followup: Using 1 dose IPV and 2 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of IPV, another sample at 3 months of age, that is one month after the first dose of IPV and just before the first dose of OPV.
  Interventions: Biological: IPV; Biological: OPV
- G2: IPV+OPV, 1 m+7d followup: Using 1 dose IPV and 2 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of IPV, another sample at 3 months and 7 days of age, that is 7 days after the first dose of OPV.
  Interventions: Biological: IPV; Biological: OPV
- G3: IPV+OPV, 2 m followup: Using 1 dose IPV and 2 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of IPV, another sample at 4 months of age, that is one month after the first dose of OPV and just before the second dose of OPV.
  Interventions: Biological: IPV; Biological: OPV
- G4: IPV+OPV, 3 m followup: Using 1 dose IPV and 2 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of IPV, another sample at 5 months of age, that is one month after the second dose of OPV.
  Interventions: Biological: IPV; Biological: OPV
- G5: OPV, 3 m followup: Using 3 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of OPV, another sample at 5 months of age, that is one month after the third dose of OPV.
  Interventions: Biological: OPV
- G6: OPV, 1 m followup: Using 3 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of OPV, another sample at 3 months of age, that is one month after the first dose of OPV and just before the second dose of OPV.
  Interventions: Biological: OPV
- G7: OPV, 1 m+7d followup: Using 3 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of OPV, another sample at 3 months and 7 days of age, that is 7 days after the second dose of OPV.
  Interventions: Biological: OPV
- G8: IPV+IPV, 1 m+7d followup: Using 2 dose IPV and 1 doses of OPV at 2, 3 and 4 months of age; Collecting two blood samples: one sample just before the first dose of IPV, another sample at 3 months and 7 days of age, that is 7 days after the second dose of IPV.
  Interventions: Biological: IPV
- G9: IPV+IPV, 2 m followup: Using 2 doses of IPV and 1 doses of OPV at 2, 3,4 months of age; Collecting two blood samples: one sample just before the first dose of IPV, another sample at 4 months of age, that is one month after the second dose of IPV and just before the first dose of OPV.
  Interventions: Biological: IPV
- G10: IPV+OPV, 1 m and 3 m followup: Using 1 dose IPV and 2 doses of OPV at 2, 3 and 4 months of age; Collecting three blood samples: one sample just before the first dose of IPV, another sample at 3 months of age, that is one month after the first dose of IPV and just before the first dose of OPV;the third sample at 5 months of age, that is one month after the second dose of OPV.
  Interventions: Biological: IPV; Biological: OPV
- G11: IPV+OPV, 1 m+7d and 2 m followup: Using 1 dose IPV and 2 doses of OPV at 2, 3 and 4 months of age; Collecting three blood samples: one sample just before the first dose of IPV, another sample at 3 months and 7 days of age, that is 7 days after the first dose of OPV,the third sample at 4 months of age, that is one month after the first dose of OPV.
  Interventions: Biological: IPV; Biological: OPV
- G12: IPV+IPV,1 m+7d and 2 m followup: Using 2 dose IPV and 1 doses of OPV at 2, 3 and 4 months of age; Collecting three blood samples: one sample just before the first dose of IPV, another sample at 3 months and 7 days of age, that is 7 days after the second dose of IPV,the third sample at 4 months of age, that is one month after the second dose of IPV.
  Interventions: Biological: IPV

INTERVENTIONS:
Biological: IPV — IPV will be vaccinated at 2 months of age act as the first dose of poliovirus vaccine in the study group1 to group 4,group8 to group 11. IPV will be given at 3 month of age act as second vaccine in group 8,9,12
  Groups: G10: IPV+OPV, 1 m and 3 m followup; G11: IPV+OPV, 1 m+7d and 2 m followup; G12: IPV+IPV,1 m+7d and 2 m followup; G1: IPV+OPV, 1 m followup; G2: IPV+OPV, 1 m+7d followup; G3: IPV+OPV, 2 m followup; G4: IPV+OPV, 3 m followup; G8: IPV+IPV, 1 m+7d followup; G9: IPV+IPV, 2 m followup
Biological: OPV — OPV will be vaccinated at 3 and 4 months of age, act as the second and third dose of poliovirus vaccine in the study group 1 to group 4,group 10 to group 11.
  OPV will be vaccinated at 2, 3 and 4 months of age act as the full three primary immunization doses of polio virus vaccine in the study group 5 to group 7.
  Groups: G10: IPV+OPV, 1 m and 3 m followup; G11: IPV+OPV, 1 m+7d and 2 m followup; G1: IPV+OPV, 1 m followup; G2: IPV+OPV, 1 m+7d followup; G3: IPV+OPV, 2 m followup; G4: IPV+OPV, 3 m followup; G5: OPV, 3 m followup; G6: OPV, 1 m followup; G7: OPV, 1 m+7d followup

SUMMARY:
The Purpose of this study is to assess the seroconversion using inactivated poliovirus vaccine (IPV) and oral poliovirus vaccine (OPV) sequential schedule in pilot areas where IPV was phased introduced into national immunization program (NIP) in China.

DETAILED DESCRIPTION:
Objective:

1. To evaluate the seroprotection rates after the 3 doses of primary polio vaccination among age eligible children in pilot areas where the IPV was introduced into NIP;
2. To evaluate the seroprotection rates after different dose(s) of polio vaccine(s) using sequential schedule.

Sample size:752

1. Jilin shall select 120 subjects to collect blood samples for evaluation of immune response,of whom 90 will be given OPV as second vaccine and 30 will be given IPV as second vaccine
2. Hubei shall select 132 subjects to collect blood samples for evaluation of immune response,of whom 102 will be given OPV as second vaccine and 30 will be given IPV as second vaccine
3. Ningxia shall select 260 subjects to collect blood samples for evaluation of immune response. The subject will be divided into 5 groups.
4. In Guangdong province,120 children will be selected as subjects , of whom 80 children will be given OPV as first vaccine and 40 children will be given IPV as first vaccine.
5. Tianjin shall select 120 subjects to collect blood samples for evaluation of immune response, of whom 80 will be given OPV as second vaccine and 30 will be given IPV as second vaccine

Organization Chart of the Study:

* Chinese Centers for Disease Control and Prevention (China CDC) lead the overall study, and be responsible for the study design, supervise the five selected provinces, conduct field monitor, data analysis and result distribution and explanation.
* The five pilot Provincial CDCs conduct the supervision and monitoring of 1-2 counties CDCs in each of pilot province.
* The County CDCs organize several vaccination clinics to recruit the subjects who meet the Inclusion criteria.

Quality Assurance Plan:

* China CDC and provincial CDC will monitor and supervise the field work, ensure the quality of the study.
* County CDCs organize vaccination clinics to service the subjects receiving timely polio vaccines in accordance with the immunization schedule, and that the blood samples are collected in accordance with the required timeline in difference groups.
* Clinic doctors will communicate and explain the purpose and procedure of the survey to parents, and the signed informed consent from by parents will be obtained before the children participate the study.
* The target drop-out rate of subjects without the second blood samples in each province should be less than 10%.
* The samples will be tested for polio antibody in a qualified laboratory, which should be a World Health Organization certified polio network laboratory in China.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children who are regular residents in the pilot counties where the immune response is evaluated in pilot provinces.
* Receiving the polio vaccination at 2, 3 and 4 months old with an interval of 28-35 days between doses according to national immunization schedule. The first dose of vaccine was administered at 2 full months old and less than 3 full months old.
* No rotavirus vaccine was administered during the period of primary polio vaccinations, and no vaccines of category 2 (private market) were administered simultaneously with polio vaccine. If vaccines of category 2 other than rotavirus vaccine were administered, they should be administered with a space of at least 2 weeks with polio vaccination.

Exclusion Criteria:

* The first dose of polio vaccine was administered at more than 3 months old regardless of the reasons.
* Children didn't get proper type and doses of vaccine as the protocal required.
* Children with known immunodeficiency conditions.
* Immunosuppressive agents or blood products were used after birth.
* Vaccine contraindications.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants will be seclected from the vaccination clinics. The study will be in five provinces, which conduct the pilot project of IPV phased introduction into national immunization program. In each province, 1-2 counties will be selected, and then selected several vaccination clinics.
Sampling Method: Non-Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | One month after the specific dose of IPV or OPV
  Calculate the percentage of subjects with seroconversion after each dose of IPV or OPV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Huaqing Wang, MD, PhD, Principal Investigator — Centers for Disease Control and Prevention, China; Zhijie An, MD, MPH, Study Director — Centers for Disease Control and Prevention, China; Zijian Feng, MD, MPH, Study Chair — Centers for Disease Control and Prevention, China
Locations (5):
- China (5):
  - Guangdong Center for Disease Control and Prevention, Guangzhou, Guangdong
  - Hubei Center for Disease Control and Prevention, Wuhan, Hubei
  - Jilin Center for Disease Control and Prevention, Changchun, Jilin
  - Ningxia Center for Disease Control and Prevention, Yinchuan, Ningxia
  - Tianjin Center for Disease Control and Prevention, Tianjin, Tianjin Municipality

REFERENCES:
- [Background] Grassly NC. Immunogenicity and effectiveness of routine immunization with 1 or 2 doses of inactivated poliovirus vaccine: systematic review and meta-analysis. J Infect Dis. 2014 Nov 1;210 Suppl 1(Suppl 1):S439-46. doi: 10.1093/infdis/jit601. Epub 2014 Mar 14. PMID 24634499
- [Background] Resik S, Tejeda A, Sutter RW, Diaz M, Sarmiento L, Alemani N, Garcia G, Fonseca M, Hung LH, Kahn AL, Burton A, Landaverde JM, Aylward RB. Priming after a fractional dose of inactivated poliovirus vaccine. N Engl J Med. 2013 Jan 31;368(5):416-24. doi: 10.1056/NEJMoa1202541. PMID 23363495